CLINICAL TRIAL: NCT02928328
Title: Vurdering af Perifere GABAA-receptorer Med Henblik på Lokal Smertelindring
Brief Title: Assessment of Peripheral GABA Receptors for Local Pain Relief
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Brian E Cairns, Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: N-20160037
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Pain
Keywords: craniofacial pain; masticatory muscle; burning mouth syndrome; temporomandibular disorders
MeSH Terms: conditions — Pain; Facial Pain; Burning Mouth Syndrome; Temporomandibular Joint Disorders | interventions — gamma-Aminobutyric Acid; Lidocaine; Capsaicin; Lorazepam; Glutamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GABA oral solution (Experimental): This study will test if oral administration of GABA containing solutions will reduce the pain and sensitivity induced by application of capsaicin to the tongue of healthy human subjects.
  Interventions: Drug: GABA oral solution
- Intramuscular GABA (Experimental): This study will test the hypothesis that intramuscular injection of GABA alone will not be painful, but will reduce muscle pain sensitivity in healthy human subjects.
  Interventions: Drug: Intramuscular GABA
- Pain modulation (Experimental): This study will test the hypothesis that intramuscular injection of GABA with glutamate will decrease the intensity of glutamate-evoked muscle pain in healthy human subjects.
  Interventions: Drug: Pain modulation

INTERVENTIONS:
Drug: GABA oral solution — Oral mouth wash containing either GABA, lidocaine or distilled water will be used to decrease burning tongue pain produced by capsaicin
  Other Names: gamma aminobutyric acid; lidocaine; distilled water; capsaicin
  Arms: GABA oral solution
Drug: Intramuscular GABA — The effect of intramuscular injection of GABA or lorazepam will be compared with buffered isotonic saline
  Other Names: gamma aminobutyric acid; lorazepam; buffered isotonic saline
  Arms: Intramuscular GABA
Drug: Pain modulation — The effect of GABA alone or in combination with lorazepam on muscle pain produced by intramuscular injection of glutamate will be assessed.
  Other Names: gamma butyric acid; glutamate; lorazepam
  Arms: Pain modulation

SUMMARY:
The effect of peripheral GABAA receptor activation on pain and sensitivity in healthy human subjects has never been investigated. However, as earlier studies suggest that activation of peripheral GABAA receptors is anti-nociceptive in rats, it is important to determine if these findings can be translated into human subjects to determine if peripheral GABAA receptors are a viable target for future analgesic drug development.

DETAILED DESCRIPTION:
Subproject I This study will test if oral administration of GABA containing solutions will reduce the pain and sensitivity induced by application of capsaicin to the tongue of healthy human subjects. Thirty, pain-free men (n=15) and women (n=15) for the oral cavity study.

Subproject II This study will test the hypothesis that intramuscular injection of GABA alone will not be painful, but will reduce muscle pain sensitivity in healthy human subjects. Thirty, pain-free men (n=15) and women (n=15) will be recruited for the intramuscular GABA injection studies

Subproject III This study will test the hypothesis that intramuscular injection of GABA with glutamate will decrease the intensity of glutamate-evoked muscle pain in healthy human subjects. Thirty, pain-free men (n=15) and women (n=15) will be recruited for the intramuscular glutamate and GABA injection studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-40 years
* Free from ongoing or chronic pain
* Adequate conversational English

Exclusion Criteria:

* Pregnancy or intent to become pregnant, breast feeding
* Signs or symptoms of any serious systemic diseases
* Current malignancies
* High blood pressure
* Requirement for chronic administration of psychiatric, analgesic or other medications that might influence their response to pain
* Frequent recreational drug or alcohol use
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Rating | continuously for 95 minutes
  visual analogue scale

SECONDARY OUTCOMES:
Jaw Function Tests | every 5 min for 50 minutes
  maximal jaw opening, maximal bite force
Quantitative Sensory testing | every 10 min for 90 min
  Pressure detection and pain threshold, thermal detection and pain threshold

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Cairns, PhD DrMed, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Y, Wang K, Arendt-Nielsen L, Cairns BE. gamma-Aminobutyric acid (GABA) oral rinse reduces capsaicin-induced burning mouth pain sensation: An experimental quantitative sensory testing study in healthy subjects. Eur J Pain. 2018 Feb;22(2):393-401. doi: 10.1002/ejp.1128. Epub 2017 Oct 11. PMID 29024230